CLINICAL TRIAL: NCT02293811
Title: Decoding of the Expression of Tumor Suppressor P2RX7 in Inflammatory and Malignant Colonic Mucosa
Acronym: P2RX7
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the tissue mass of each biopsy sample was not sufficient to perform an exploratory analysis to assess the level of expression of the P2RX7 protein.
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-AOI-04
Record Dates: First submitted 2014-11-14; First posted 2014-11-18 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Crohn Disease-Associated Colorectal Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- biopsy (Other): We will use colonic biopsies performed in the gastroenterology after obtaining consent from the patient and the agreement of the committee for the protection of persons. 5 biopsy will be performed for all patients except those with colon cancer for xhich we realize only 3 colonic biopsy (1 in healthy area and 2 in cancerous area )
  To obtain statistically significant results we will establish the following six study groups, as far as possible matched for age and sex:
  * healthy patients;
  * patients with colonic Crohn disease in acute phase;
  * patients with colonic Crohn disease in chronic phase;
  * patients with ulcerative colitis in acute phase;
  * patients with ulcerative colitis in chronic phase;
  * patients with colon cancer
  Interventions: Other: Analysis

INTERVENTIONS:
Other: Analysis — An additional blood sample (10ml) will be taken on the day of hospitalization to achieve the genomic studies in search of mutations in constitutional DNA of circulating lymphocytes and acquired mutations of DNA circulating.
  We will use the technique of tissue-microarray to analyze the expression level of P2RX7 both in epithelial cells than in stromal cells inflammatory.
  Genotyping will be conducted partly on colonic biopsies and also on blood samples (to demonstrate the feasibility of this technique much less debilitating).

SUMMARY:
The inflammatory tumor micro-environment is a consequence and a driver of tumorogenesis. On one hand it promotes antitumor immune responses and on the other hand it favors development and progression of cancerous lesions.

Factors regulating the complex interplay between epithelial and immune cells are still poorly characterized. Extracellular ATP (eATP) acting on the purinergic P2X7 receptors (P2RX7) has recently emerged as a key signaling pathway in the immune response.

Recent data have revealed the crucial role of P2RX7-NLRP3-Caspase-1 for priming dendritic cells (DC) within the tumor microenvironment upon treatment with certain types of chemotherapy drugs. Despite this important discovery, no previous study has so far investigated the global in vivo effect of P2RX7 modulation in inflammation-induced carcinogenesis of mucosal tissues.

Our consortium, endowed by a long standing experience in the field of mucosal immunology, inflammation and signaling, already demonstrated that the P2RX7 is differentially expressed in the mucosa of patients with active and quiescent inflammatory bowel disease (IBD), where eATP is present at very high concentration, and that P2RX7 controls an amplification loop of the inflammatory response (Cesaro et al., 2010). Furthermore, we uncovered that P2RX7 controls homeostasis, survival and function of regulatory T cells (Hubert et al., 2010). In addition, our recent demonstration that P2RX7 deficiency lowered mucosal inflammation but unexpectedly enhanced tumor formation in vivo warrants additional efforts to explore the molecular and cellular mechanisms accounting for this effect and suggest that enhancing P2RX7 function may have an anti-tumor therapeutic effect.

These observations emphasize the tumor suppressor role of P2X7 receptor, warrant further investigation to better understand the molecular mechanisms responsible for this anti-tumor effect and suggest that enhancing the function of P2X7R could have a therapeutic effect significant antitumor.

Our main objectives is to explore the role of P2RX7 in healthy, inflammatory and cancerous colonic mucosa. For this we will map the expression of the protein P2RX7 and realize genotype of P2RX7 forms in inflammatory diseases and cancer of the colon.

ELIGIBILITY:
Inclusion Criteria:

* · All the patients requiring an endoscopy within the framework of a colorectal cancer

  * All the patients requiring a low digestive endoscopy within the framework of the diagnosis or of the follow-up of a colorectal cancer, realized in the CHU of Nice.
  * Realization of a preliminary medical examination
  * Obligation for all the patients to be affiliated to the Social Security
  * Signature of the informed consent

Exclusion Criteria:

* • Pushed acute severe of the disease defined by the score of Truelove and Witss or the score of Lichtiger > 10 (cf appendix)

  * severe endoscopic Hurts returning the practice of dangerous additional biopsies
  * Disorders of the coagulation or the patient under anti-vitamin K, aspirin or clopidogrel.
  * Patient presenting an unchecked renal, respiratory, hepatic or cardiac insufficiency
  * Patient known positive HIV
  * vulnerable People: pregnant or breast-feeding women (a pregnancy test will be realized), minors, adults under guardianship or guardianships, deprived of freedom

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-02-09 (Actual); Primary Completion 2015-10-15 (Actual); Study Completion 2015-12-15 (Actual)

PRIMARY OUTCOMES:
Analysis of expression of P2RX7 | One time
  The evaluation of the level of expression of P2RX7 will realized by tissue microarray (TMA). TMA is produced using colonic biopsies fixed in 10% formalin. Plug of paraffin embedded tissue will be selected from stained with hematoxylin eosin saffron corresponding cuts. This selection of the tissue area taken from the donor block must be done carefully, conditioning the quality of the "array". In practice, for each patient, 3 Plug of 0.6 mm shall be taken from a biopsy performed in pathological tissue. A total of 156 spots TMA of 0.6 mm diameter plug shall be included according to a pre-established in a receiver block plane (consisting of virgin paraffin).

SECONDARY OUTCOMES:
Five isoforms of the P2RX7 protein | one time
  Five isoforms of the P2RX7 protein are described and each of its isoforms have many single nucleotide polymorphisms (SNPs). Among the 1754 mutations identified, 33 have been referenced in Pubmed publications and 4 are associated with diseases such as osteoarthritis, chronic pain and leukemias. Thus, the function of P2X7R may be affected by the expression of variants "gain of function" or "loss of function" and it is important to map the expression of these variants to anderstand the role of P2X7R in inflammatory bowel diseases and colonic cancer.
  Genotyping will be conducted on colonic biopsy and on blood samples (to demonstrate the feasibility of this technique much less debilitating). We will use the platform MassARRAY SNP multiplex (present in my home lab) by following the procedures established by the platform.

CONTACTS AND LOCATIONS:
Overall Officials: HEBUTERNE Xavier, PhD, Principal Investigator — CHU de Nice, Hôpital Archet, Gastroentérologie
Locations (1):
- CHU de Nice, Nice, Alpes-Maritimes, France